CLINICAL TRIAL: NCT02082873
Title: A Prospective Trial of Nonconvulsive Electrographic Seizure Detection by Nurses in the Adult Neuro ICU Using a Panel of Quantitative EEG Trends
Brief Title: Nonconvulsive Seizure Identification on Quantitative EEG by Neuro ICU Nurses
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00052133
Record Dates: First submitted 2014-03-05; First posted 2014-03-10 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-04

CONDITIONS: Nonconvulsive Seizures
Keywords: Quantitative EEG; Nonconvulsive seizures; ICU EEG monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research is being conducted to determine if Neuroscience intensive care unit (ICU) nurses are able to identify seizures by reviewing quantitative EEG (qEEG) that is running at the bedside. QEEG is the application of mathematical and analytical techniques to analyze EEG signals. Several hours of data can be displayed on a single screen in several graphical panels. Routine evaluation of EEG data consists of manual inspection of each page of EEG data by a trained neurophysiologist (a neuro ICU doctor) and can be quite time-consuming. In most cases, this data can only be reviewed intermittently and interpretation is almost always relayed to the primary clinical team after the seizures have occurred. Theoretically,qEEG graphical displays can provide a simplified view of complex EEG data that could possibly be used by non-neurophysiologists, such as Neuro ICU nurses. Our hypothesis is that Neuro ICU nurses are able to accurately identify recurrent seizures in real-time.

DETAILED DESCRIPTION:
PROTOCOL TITLE A prospective trial of nonconvulsive electrographic seizure detection by nurses in the adult Neuro ICU using a panel of quantitative EEG trends

PURPOSE OF STUDY The primary objective of this prospective study is to determine the sensitivity and specificity of quantitative EEG (qEEG) trends in the identification of recurrent nonconvulsive electrographic seizures by non-neurophysiologists in adult patients admitted to the Duke Neuro Intensive Care Unit (Neuro ICU). Our hypothesis is that bedside Neuro ICU nurses using a panel of qEEG trends can identify recurrent nonconvulsive seizures (NCS) with adequate sensitivity and specificity.

Secondary objectives include identifying seizure and EEG characteristics that make NCS more or less likely to be detected on qEEG. These characteristics include average seizure duration, spatial extent of the seizure (focal, hemispheric or bilateral/generalized) and the EEG background (periodic vs. non-periodic and epileptiform vs. non-epileptiform).

PRINCIPLE INVESTIGATOR Dr. Saurabh R. Sinha MD, will be the principal investigator (PI) on this project and is responsible for the study design, generation and analysis of data, presentation of reports, and protection of human subjects in the performance of the clinical investigation. His contact information is provided below.

Saurabh R. Sinha, M.D. 295 Hanes House, 330 Trent Drive. Box 102350 Duke University Medical Center. Durham, NC 27710. Phone: 919-684-8485. Fax: 919-684-8955. Email: saurabh.sinha@duke.edu

BACKGROUND AND SIGNIFICANCE

Due to the increased awareness of nonconvulsive seizures (NCS) and nonconvulsive status epilepticus (NCSE) in patients admitted to the NICU, the utilization of continuous EEG (cEEG) monitoring in the NICU is rising. qEEG is a potential tool that can aid in the interpretation of large volumes of EEG data. qEEG is the application of mathematical and analytical techniques to characterize and analyze EEG signals. Several hours of data can be displayed on a single screen in several graphical panels. Routine evaluation of EEG data consists of manual inspection of each page of EEG data and can be quite time-consuming. Since continuous review of EEG data is not possible, EEG data is always relayed to the primary clinical team in a post-hoc manner which is not ideal. Theoretically, qEEG graphical displays can provide a simplified view of complex EEG data that could possibly be used by non-neurophysiologists, such as Neuro ICU nurses.

There have been no studies in the adult or pediatric population that have prospectively evaluated the use of qEEG by non-neurophysiologists to identify recurrent NCS. Given that our retrospective data show that neurophysiologists and non-neurophysiologists have similar sensitivity and specificity in identifying the presence of NCS on qEEG panels, our hypothesis is that Neuro-ICU nurses will have an acceptable sensitivity and specificity in prospectively identifying recurrent NCS.

DESIGN AND PROCEDURES

This is an observational, prospective evaluation of Neuro ICU nurses' ability to detect NCS via qEEG running at the bedside. The study will not affect clinical management decisions or patient care. It will utilize DUHS Neuro ICU nurses that will serve as qEEG readers.

The goal of this study is to compare the accuracy of Neuro-ICU nurses' ability to detect NCS on bedside qEEG and post hoc review of the corresponding raw EEG by blinded, board-certified neurophysiologists. The neurophysiologists are blinded to the Neuro ICU nurses prospective seizure identification.

We plan to enroll a sample of 40 nurses and 30 adult patients who are already on continuous video electroencephalogram (EEG) monitoring during their admission to the Duke Neuroscience ICU. In this prospective study we will include adults who are clinically suspected to have NCS, defined by the fact that the treatment team physician has requested cEEG monitoring. The treating physician will make the decision to initiate cEEG monitoring and determine the duration of monitoring. We will exclude subjects with convulsive seizures without concern for NCS.

All eligible subjects will be consented for enrollment after the clinical team has decided that the patient will be placed on cEEG monitoring. Subsequently, the neurophysiology fellow will review the raw EEG intermittently as this is the standard of care. Once the neurophysiology fellow has detected NCS, the research team will be contacted by either the clinical Neuro ICU team or the neurophysiology team if the patient is deemed appropriate to continue participation in the study.

Nurses will be consented for their participation in the trial as it involves their ability to detect NCS with the use of bedside qEEG trends. Neuro ICU nurses who consent will receive training on qEEG monitoring by the research team via a 15 minute online PowerPoint presentation. In addition, a binder containing printouts of the training PowerPoint presentation will be attached to each EEG machine.

A single printout of a qEEG panel, containing the sentinel seizure captured on cEEG monitoring will be displayed next to the cEEG machine. The NCS will be clearly marked by the research team. All patients undergoing cEEG monitoring at Duke have qEEG running simultaneously in addition to the raw EEG. The program that creates the qEEG display is Magic Marker developed by Persyt, Inc. Neuro ICU nurses will be asked to check the qEEG screen hourly and record the number of seizures (similar in appearance to the sentinel seizure qEEG print out) seen on the qEEG display. A 24 hour log will be attached to the EEG machine. If a patient and a nurse are enrolled in the study, but the second nurse on the later shift has not agreed to participate in the trial then we will either end the study or ask the second nurse if he/she would like to participate. There are nurses from the float pool that may be interested, and if so, we will provide a one-on-one training session at the beginning of their shift and consent them. At one hour intervals the nurse will mark one of the following options: no seizures, 1-2 seizures, 3-5 seizures, 6-10 seizures or >10 seizures. The absolute times that the nurse should evaluate the qEEG display will be determined by the study team at the time of enrollment and clearly marked on the log sheet. The standard of practice of the neurophysiology fellow independently reviewing the raw EEG intermittently will continue unchanged. Treatment of recurrent NCS will be at the discretion of the Neuro ICU team in conjunction with the neurophysiology team. The nurse's review of the qEEG will have no impact on patient care or treatment decisions.

The nurse will review the subject's qEEG for the duration of their shift (12 hours) or for only part of their shift. The total duration of the study will be for 24 hours or when the treating physician discontinues continuous EEG monitoring, whichever is shorter. If the first nurse participates in the study, but the nurse on the second shift has not agreed to participate, then the study will stopped.

After completing enrollment, the qEEG data and raw EEG data will be de-identified by study author (CW). Board-certified neurophysiologists and study authors (SS and CS) will review the raw EEG data independently to identify seizures. Electrographic seizures will be identified using published criteria [15]. In the case of discrepancy in the identification of seizures the two authors will review the studies together and establish a consensus. Each hour of raw EEG will be placed into the follow categories: no seizures, 1-2 seizure, 3-5 seizures, 6-10 seizures or >10 seizures. In addition, the average seizure duration, the spatial extent of each seizures (focal, hemispheric or generalized/bilateral), and primary background EEG abnormalities will be determined by the author and board-certified neurophysiologist, CS, from the raw EEG.

SELECTION OF SUBJECTS

Neuroscience ICU Nurses:

All Neuroscience ICU nurses will be asked to participate.

Subjects:

The responsible treating team in the Adult Neuro ICU will identify subjects after the treating physician has decided to initiate cEEG monitoring. No restrictions are made with regard to gender, race, religion or underlying cause for hospitalization, including prior history of seizure disorder.

SUBJECT RECRUITMENT AND COMPENSATION Appropriate subjects will be identified by the treating team in the Adult Neuro ICU. It will be at the sole discretion of the treating team in the Adult Neuro ICU or the clinical neurophysiology team to notify a research coordinator to approach the patient for recruitment into the study. Subject demographics will mirror that of the patient demographics of the Duke Adult Neuro ICU. No compensation will be provided.

CONSENT PROCESS

Neuroscience ICU Nurses:

The study will be introduced to all Neuro ICU nurses via an email request to participate in the study. The consent form will be reviewed with all nurses willing to participate in the trial. The study physicians will review the consent forms individually with each nurse in the Duke Medical Pavilion conference room and answer any questions individually at that time. Those that agree to participate in the study and sign the consent form will attend a brief, 15 minute training session on qEEG monitoring presented by the study authors (SS, CS and CW). Their participation is completely voluntary and their recorded responses of qEEG interpretation will be used as part of the project data. No identifying information will be recorded. It will be made explicitly clear that there will be no penalty for not participating and that no incentives will be provided.

Subjects and Subjects Legal Representative:

The study will be introduced to the patient or Legally Authorized Representative (LAR) by a member of the clinical team. If the patient or LAR is willing to participate, the study team will approach them. Informed consent will be obtained by the PI, Study Coordinator, or other Key personnel for all subjects in the study. Consent will be obtained from the patient or LAR, as defined by Duke guidelines, if the patient is unable to provide consent. The patient will be assessed for impaired decision-making at the time of consent. All patients requiring cEEG monitoring will require involvement of a neurologist who will determine the ability to consent if that determination has not already been made either by the PI or other investigators on the trial. All investigator personnel on this trial are neurologists. Consent will be obtained in a quiet, private location to protect the privacy of the prospective participant. Potential participants will be identified by bedside evaluation at DUHS Neuro ICU. Once the participant is identified, the patient and/or family will be notified of the opportunity to participate in the project, and the purpose of the study will be reviewed in addition to all of the risks and benefits of participation. The entire consent form will be reviewed and all questions will be addressed. It will be made explicitly clear to all participants and LARs that no additional procedures will be performed as part of this trial and that no incentives will be provided.

SUBJECT'S CAPACITY TO GIVE LEGALLY EFFECTIVE CONSENT Many subjects will not have the capacity to provide consent given the nature of the study and acuity of the disease. Consent will be obtained from the subject's legal representative. Periodic assessment of capacity will be assessed by the research coordinator, and if deemed to have capacity the subject will be presented with the opportunity to be consented.

STUDY INTERVENTIONS The standard of care will continue unchanged, and this consists of intermittent raw EEG review by the neurophysiology team. No interventions will come to the participating subject based on qEEG data review by the Neuro ICU nurses, but rather will continue to rely on the current standard of care with the existing infrastructure using raw EEG. All decisions to treat NCS will be at the sole discretion of the treating team and responsible care physicians. The duration of continuous EEG monitoring will be determined solely by the treating team or responsible care physician.

RISK/BENEFIT ASSESSMENT

Subjects and Subjects Legal Representative:

There are no physical, psychological, legal, or economic risks identified. Social risks include the decision to choose to participate or not participate. Cognitively impaired adults may be recruited as subjects given the acuity and sequela of NCS. Special precautions include the deferring to the subjects legal representative for consent in this situation. Should the subject or subjects LAR choose not to participate there will be no repercussions and medical care will continue per the treating team. There will be no direct benefit to the patients enrolled in the study.

Neuroscience ICU Nurses:

There are no physical or psychological risks identified. The nurse's decision to participate or not will not have repercussions. The decision to participate will have no ramifications on employment status with Duke University Hospital (job classification, pay, etc.). The neuroscience ICU nurses will benefit from the study by receiving training on qEEG interpretation.

COSTS TO THE SUBJECTS

Subjects and Subjects Legal Representative:

There will be no additional costs that the patient's will incur as a result of participation.

Neuroscience ICU Nurses:

There will be no costs that the Neuro ICU nurses will incur as a result of participation.

DATA ANALYSIS AND STATISTICAL CONSIDERATIONS We will determine the sensitivity and specificity of the use of qEEG trends by Neuro ICU nurses in identifying recurrent nonconvulsive seizures in critically ill patients with acute or chronic neurologic injuries. This will be calculated by comparing the number of suspected seizures marked by Neuro ICU nurses via qEEG displays to the number of seizures identified by the gold standard analysis of the raw EEG.

Standard test characteristics (sensitivity, specificity, positive predictive value and negative predictive value, positive likelihood ratio and negative likelihood ratio) will be calculated for the ability to detect the presence or absence of seizures. Contingency analysis will be used to make several comparisons of the mean diagnostic accuracy of the Neuro ICU nurses: 1. short (< 25th percentile) vs. long (> 75th percentile) seizures; 2. spatial extent of seizures (generalized vs. hemispheric vs. focal); 3. Background EEG pattern (epileptiform vs. non-epileptiform and periodic vs. non-periodic). The chi-square statistic will be calculated for each these analyses. For all calculations, a p-value < 0.05 will be considered statistically significant.

DATA AND SAFETY MONITORING Raw and qEEG data will be obtained and stored (as it is currently). The qEEG and raw EEG data will be anonymized after the subject has completed participation in the study. Although all EEG data in the Neuro ICU is recorded with video for clinical purposes, no video will be retained during this project. The anonymized data will be used solely by research investigators.

Standard clinical practice will not be altered during this study. There should be no impact on patient care.

PRIVACY, DATA STORAGE AND CONFIDENTIALITY

Data to be collected will include the digital EEG portion of our cEEG monitoring records and their corresponding qEEG panels. Although all EEG data in the Neuro ICU is recorded with video for clinical purposes, no video will be retained during this project. After extracting the relevant data from the complete cEEG file, all identifying information will be removed and the EEG will be numerically indexed in the data set. All cEEG and qEEG data is currently collected locally (bedside PC) on the monitoring system and automatically copied to the central server for remote review. Once the data is collected, the files are centrally reviewed, and at that point can be copied to the project computer for indexing, extraction of segments and de-identification of the data. All PHI data will be removed leaving no record of the origin of the data. Clinical data will be stored on the Duke IT maintained network server. The de-identified cEEG and qEEG data will be stored on the Isilon storage server behind Duke's firewall. The de-identified cEEG or qEEG data will not be shared with any parties outside Duke.

Clinical data will be collected from the Duke electronic medical record system. This includes age, race, gender, primary diagnosis, and reason of cEEG monitoring. As part of the study protocol, no PHI will be recorded at any time. PHI will only be reviewed to extract relevant study information, such as patient demographics and official interpretation of the cEEG by the neurophysiology team. This review process will occur less than 24 hours after study initiation. After the relevant information is extracted, the demographic data, cEEG data and qEEG data will be anonymized.

Research data will be stored on a Duke IT maintained network server. Confidentiality will be ensured as no PHI or video data will be retained on this server. The de-identified cEEG and qEEG data will be used solely by research investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or older at time of consent
2. Patients undergoing cEEG monitoring to evaluate for the presence of NCS
3. Admission or pending transfer to the adult Neuro ICU
4. Informed consent by patient or patient's legally authorized representative (LAR)
5. One or more NCS identified on cEEG monitoring, confirmed by the clinical neurophysiology team

Exclusion Criteria:

1. Anticipated discharge from NICU < 24 hours
2. Anticipated duration of cEEG monitoring < 24 hours
3. Suspected diagnosis of brain death
4. Open head wound or bandage preventing application of majority of EEG electrodes
5. Treating physician deems not appropriate for subject participation
6. Seizures lasting more than 1 hour in duration
7. Convulsive seizures without concern for NCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 NeuroICU patients and 40 NeuroICU nurses
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of nurses ability to detect recurrent NCS on QEEG | within 3 months after patient enrollment
  Neuro ICU nurses will be asked to check the qEEG screen hourly and record the number of seizures (similar in appearance to the sentinel seizure qEEG print out) seen on the qEEG display. At one hour intervals the nurse will mark one of the following options: no seizures, 1-2 seizures, 3-5 seizures, 6-10 seizures or >10 seizures. The total duration of the study will be for 24 hours or when the treating physician discontinues continuous EEG monitoring, whichever is shorter.
  After completing enrollment, board-certified neurophysiologists and study authors (SS and CS) will review the raw EEG data independently to identify seizures. Each hour of raw EEG will be placed into the follow categories: no seizures, 1-2 seizure, 3-5 seizures, 6-10 seizures or >10 seizures. Standard test characteristics (sensitivity, specificity, ect) will be calculated comparing the nurses responses to the gold standard of raw EEG review.

SECONDARY OUTCOMES:
Specificity of nurses ability to detect recurrent NCS on QEEG | Within 3 months of patient enrollment
  Neuro ICU nurses will be asked to check the qEEG screen hourly and record the number of seizures (similar in appearance to the sentinel seizure qEEG print out) seen on the qEEG display. At one hour intervals the nurse will mark one of the following options: no seizures, 1-2 seizures, 3-5 seizures, 6-10 seizures or >10 seizures. The total duration of the study will be for 24 hours or when the treating physician discontinues continuous EEG monitoring, whichever is shorter.
  After completing enrollment, board-certified neurophysiologists and study authors (SS and CS) will review the raw EEG data independently to identify seizures. Each hour of raw EEG will be placed into the follow categories: no seizures, 1-2 seizure, 3-5 seizures, 6-10 seizures or >10 seizures. Standard test characteristics (sensitivity, specificity, ect) will be calculated comparing the nurses responses to the gold standard of raw EEG review.

CONTACTS AND LOCATIONS:
Overall Officials: Christa Swisher, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Claassen J, Jette N, Chum F, Green R, Schmidt M, Choi H, Jirsch J, Frontera JA, Connolly ES, Emerson RG, Mayer SA, Hirsch LJ. Electrographic seizures and periodic discharges after intracerebral hemorrhage. Neurology. 2007 Sep 25;69(13):1356-65. doi: 10.1212/01.wnl.0000281664.02615.6c. PMID 17893296
- [Background] Claassen J, Mayer SA, Kowalski RG, Emerson RG, Hirsch LJ. Detection of electrographic seizures with continuous EEG monitoring in critically ill patients. Neurology. 2004 May 25;62(10):1743-8. doi: 10.1212/01.wnl.0000125184.88797.62. PMID 15159471
- [Background] DeLorenzo RJ, Waterhouse EJ, Towne AR, Boggs JG, Ko D, DeLorenzo GA, Brown A, Garnett L. Persistent nonconvulsive status epilepticus after the control of convulsive status epilepticus. Epilepsia. 1998 Aug;39(8):833-40. doi: 10.1111/j.1528-1157.1998.tb01177.x. PMID 9701373
- [Background] Jordan KG. Neurophysiologic monitoring in the neuroscience intensive care unit. Neurol Clin. 1995 Aug;13(3):579-626. PMID 7476820
- [Background] Oddo M, Carrera E, Claassen J, Mayer SA, Hirsch LJ. Continuous electroencephalography in the medical intensive care unit. Crit Care Med. 2009 Jun;37(6):2051-6. doi: 10.1097/CCM.0b013e3181a00604. PMID 19384197
- [Background] Privitera M, Hoffman M, Moore JL, Jester D. EEG detection of nontonic-clonic status epilepticus in patients with altered consciousness. Epilepsy Res. 1994 Jun;18(2):155-66. doi: 10.1016/0920-1211(94)90008-6. PMID 7957038
- [Background] Towne AR, Waterhouse EJ, Boggs JG, Garnett LK, Brown AJ, Smith JR Jr, DeLorenzo RJ. Prevalence of nonconvulsive status epilepticus in comatose patients. Neurology. 2000 Jan 25;54(2):340-5. doi: 10.1212/wnl.54.2.340. PMID 10668693
- [Background] Vespa PM, Nuwer MR, Nenov V, Ronne-Engstrom E, Hovda DA, Bergsneider M, Kelly DF, Martin NA, Becker DP. Increased incidence and impact of nonconvulsive and convulsive seizures after traumatic brain injury as detected by continuous electroencephalographic monitoring. J Neurosurg. 1999 Nov;91(5):750-60. doi: 10.3171/jns.1999.91.5.0750. PMID 10541231
- [Background] Vespa PM, O'Phelan K, Shah M, Mirabelli J, Starkman S, Kidwell C, Saver J, Nuwer MR, Frazee JG, McArthur DA, Martin NA. Acute seizures after intracerebral hemorrhage: a factor in progressive midline shift and outcome. Neurology. 2003 May 13;60(9):1441-6. doi: 10.1212/01.wnl.0000063316.47591.b4. PMID 12743228
- [Background] Young GB, Jordan KG, Doig GS. An assessment of nonconvulsive seizures in the intensive care unit using continuous EEG monitoring: an investigation of variables associated with mortality. Neurology. 1996 Jul;47(1):83-9. doi: 10.1212/wnl.47.1.83. PMID 8710130
- [Background] Kuhlmann L, Burkitt AN, Cook MJ, Fuller K, Grayden DB, Seiderer L, Mareels IM. Seizure detection using seizure probability estimation: comparison of features used to detect seizures. Ann Biomed Eng. 2009 Oct;37(10):2129-45. doi: 10.1007/s10439-009-9755-5. Epub 2009 Jul 10. PMID 19590961
- [Background] Chong DJ, Hirsch LJ. Which EEG patterns warrant treatment in the critically ill? Reviewing the evidence for treatment of periodic epileptiform discharges and related patterns. J Clin Neurophysiol. 2005 Apr;22(2):79-91. doi: 10.1097/01.wnp.0000158699.78529.af. PMID 15805807
- [Result] Kang JH, Sherill GC, Sinha SR, Swisher CB. A Trial of Real-Time Electrographic Seizure Detection by Neuro-ICU Nurses Using a Panel of Quantitative EEG Trends. Neurocrit Care. 2019 Oct;31(2):312-320. doi: 10.1007/s12028-019-00673-z. PMID 30788707
- [Derived] Kaleem S, Kang JH, Sahgal A, Hernandez CE, Sinha SR, Swisher CB. Electrographic Seizure Detection by Neuroscience Intensive Care Unit Nurses via Bedside Real-Time Quantitative EEG. Neurol Clin Pract. 2021 Oct;11(5):420-428. doi: 10.1212/CPJ.0000000000001107. PMID 34840869